CLINICAL TRIAL: NCT05769465
Title: MAP THE SMA: a Machine-learning Based Algorithm to Predict THErapeutic Response in Spinal Muscular Atrophy
Acronym: MAP_THE_SMA-01
Status: Recruiting | Type: Observational
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Sponsor
Other Study IDs: 5488; GR-2021-12374579 (Other Grant/Funding Number: Italian Health Ministry)
Record Dates: First submitted 2023-03-03; First posted 2023-03-15 (Actual); Last update posted 2023-09-13 (Actual); Status verified 2023-03

CONDITIONS: Spinal Muscular Atrophy
MeSH Terms: conditions — Muscular Atrophy, Spinal

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (4):
- Patients treated with nusinersen
  Interventions: Drug: disease modifying treatments
- Patients treated with risdiplam
  Interventions: Drug: disease modifying treatments
- Patients treated with onasemnogene abeparvovec
  Interventions: Drug: disease modifying treatments
- Patients naive from disease modifying treatments

INTERVENTIONS:
Drug: disease modifying treatments — Patients will be enrolled if exposed to nusinersen, risdiplam, onasemnogene abeparvovec
  Groups: Patients treated with nusinersen; Patients treated with onasemnogene abeparvovec; Patients treated with risdiplam

SUMMARY:
Spinal Muscular Atrophy (SMA) is caused by the homozygous loss of the Survival Motor Neuron (SMN) 1 gene, which leads to degeneration of spinal alpha-motor neurons and muscle atrophy. Three treatments have been approved for SMA but the available data show interpatient variability in therapy response and, to date, individual factors such as age or SMN2 copies,cannot fully explain this variance.

The aim of this project is:

* collect clinical data and patient-reported outcome measures (PROM) from patients treated with nusinersen, risdiplam, onasemnogene abeparvovec,
* identify novel biomarkers and RNA molecular signature profiling,
* develop a predictive algorithm using artificial intelligence (AI) methodologies based on machine learning (ML), able to integrate clinical outcomes, patients' characteristics, and specific biomarkers.

This effort will help to better stratify the SMA patients and to predict their therapeutic outcome, thus to address patients towards personalized therapies.

ELIGIBILITY:
Inclusion Criteria:

* confirmed genetic diagnosis of SMA (5q)
* clinical phenotype of type I or II or III;
* able to provide (patient/caregiver) written informed consent

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients cared for at Policlinico Gemelli with confirmed genetic diagnosis of SMA (5q) type I or II or III; written informed consent obtained from the participants or their families.
Sampling Method: Non-Probability Sample
Enrollment: 247 (Estimated)
Dates: Start 2023-04-01 (Actual); Primary Completion 2025-11-01 (Estimated); Study Completion 2026-04-01 (Estimated)

PRIMARY OUTCOMES:
Collect clinical data and patient-reported outcome measures (PROM) from patients treated with nusinersen, risdiplam, onasemnogene abeparvovec | 30 months
Identify novel biomarkers and RNA molecular signature profiling | 30 months
Develop a predictive algorithm using artificial intelligence (AI) methodologies based on machine learning (ML), able to integrate clinical outcomes, patients' characteristics, and specific biomarkers | 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Giorgia Coratti, PhD, Principal Investigator — Fondazione Policlinico Universitario Agostino Gemelli IRCCS
Locations (1):
- Fondazione Policlinico Universitario Agostino Gemelli IRCCS, Roma, Italy